CLINICAL TRIAL: NCT01580748
Title: Phase2, Single Group, Open Clinical Trial to Evaluate the Efficacy and Safety of Roflumilast in Symptomatic Bronchiectasis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hoil Yoon, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-1109-066-002
Record Dates: First submitted 2012-04-18; First posted 2012-04-19 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Symptomatic Bronchiectasis
MeSH Terms: interventions — Roflumilast

ARMS (1):
- Treatment arm (Experimental): single arm study
  Interventions: Drug: Roflumilast

INTERVENTIONS:
Drug: Roflumilast — 500 microgram once daily for 16 weeks

SUMMARY:
There is currently no effective treatment of bronchiectasis other than treating its complications such as infection, bleeding, etc. Roflumilast is a newly developed anti-inflammatory drug that has proven to be effective in stable COPD. We hypothesized that Roflumilast might be effective in symptomatic bronchiectasis patients

ELIGIBILITY:
Inclusion Criteria:

* Bronchiectasis on CT
* chronic (>3 months) cough or sputum

Exclusion Criteria:

* needs hospitalization
* life expectancy of less than six months
* pregnancy or breast feeding
* history of acute respiratory infection within 4 weeks
* history of taking antibiotics within 4 weeks
* active hemoptysis
* %predicted FEV < 30%
* severe liver disease (Child Pugh Class B or C)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
change of CASA-Q score | 16 weeks

SECONDARY OUTCOMES:
change of FEV1 | 16 weeks
change of FVC | 16 weeks
alanine transaminase | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyeongi-do, South Korea